CLINICAL TRIAL: NCT06373575
Title: Inferior Vena Cava and Lung Ultrasound B-lines Guided Decongestion in Critically Ill Kidney Failure Patients With Heart Failure: a Single-center, Prospective, Randomized Controlled Intervention Study
Brief Title: IVC and Lung Ultrasound B-lines Guided Decongestion in Critically Ill ESKD Patients With Heart Failure
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-SR-891
Record Dates: First submitted 2024-04-10; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: End-stage Renal Disease
Keywords: Kidney Failure, Chronic; heart failure
MeSH Terms: conditions — Kidney Failure, Chronic; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Fluid removal with the guidance of lung and inferior vena cava ultrasound before prolonged hemodialysis
  Interventions: Procedure: Lung and inferior vena cava ultrasound guidance
- Control group (Active Comparator): Fluid removal with the conventional protocol
  Interventions: Procedure: Conventional protocol guidance

INTERVENTIONS:
Procedure: Lung and inferior vena cava ultrasound guidance — The lung and inferior vena cava ultrasound will be utilized as guidance for the development of a dialysis prescription for prolonged hemodialysis.
  Arms: Intervention group
Procedure: Conventional protocol guidance — Fluid removal using conventional protocol including blood pressure and physical examination
  Arms: Control group

SUMMARY:
The objectives of this trial are to determine whether, in critically ill ESKD patients randomization to fluid removal guided by lung and inferior vena cava ultrasound, compared to standard care, leads to Improved pulmonary congestion (primary outcome); and safety (secondary outcome) in the short-term.

DETAILED DESCRIPTION:
The point-of-care ultrasound was thought useful in the management of fluid in critically ill patients. At present, the role of the lung and inferior vena cava ultrasound is unclear in the management of decongestion of heart failure in kidney failure (KF) patients using prolonged hemodialysis. The investigators aim to explore the effect of pre-dialysis probing with the lung and inferior vena cava to guide fluid removal as compared with conventional protocols on the improvement of heart failure symptoms in patients with KF with heart failure under prolonged hemodialysis in the short-term.

ELIGIBILITY:
Inclusion Criteria:

1. patients meet the diagnostic criteria for end-stage renal disease;
2. indications that the patient may be experiencing signs and/or symptoms of heart failure, and based on the serum N-terminal pro-brain natriuretic peptide level of greater than 11,215. 2 ng/L;
3. patients may require prolonged intermittent renal replacement therapy due to volume overload;
4. patients ≥18 yo and ≤80 yo;
5. either the patient or a family member signs the informed consent;
6. patients will undergo at least two sessions of prolonged hemodialysis.

Exclusion Criteria:

1. history of malignancy or psychiatric disease;
2. patients with a history of congenital heart disease or hypertrophic cardiomyopathy;
3. coagulation abnormalities, intracranial, visceral or gastrointestinal bleeding in the past 3 months, or contraindications to heparin anticoagulation;
4. The duration of prolonged hemodialysis <8 hours;
5. Ultrasound unable to monitor the inferior vena cava, or can't access the date;
6. Pregnancy;
7. Patients with severe respiratory failure;
8. Patients with combined severe infections, such as patients with sepsis;
9. Presence of pre-dialysis hypotension: systolic blood pressure <90 mmHg;
10. other conditions deemed ineligible by physicians.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in pulmonary congestion score | within 72 hours following randomization
Improvement in heart failure symptoms score | within 72 hours following randomization

SECONDARY OUTCOMES:
Total ultrafiltration volume | within 72 hours following randomization
Mean ultrafiltration rate during prolonged hemodialysis | within 72 hours following randomization
Fluid balance (total outflow - total inflow) | within 72 hours following randomization
Lung B-line reduction | within 72 hours following randomization
The change of width of inferior vena cava | within 72 hours following randomization
Incidence of hypotension during prolonged hemodialysis | within 72 hours following randomization
Blood pressure variability during the prolonged hemodialysis | within 72 hours following randomization
In-hospital mortality | From date of randomization until the date of discharge or date of death from any cause, whichever came first, assessed up to 100 days
Length of hospital stay | From date of randomization until the date of discharge or date of death from any cause, whichever came first, assessed up to 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Buyun Wu, PhD, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No